CLINICAL TRIAL: NCT03423082
Title: Pilot Study to Assess the Potential Clinical Utility of 18F Fluciclovine PET for Cervical and Endometrial Cancer Compared With 18F FDG PET
Brief Title: Pilot Study to Assess the Potential Clinical Utility of 18F Fluciclovine PET for Cervical and Endometrial Cancer.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Limited subject enrollment
Sponsor: Nghi Nguyen (Other)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Sponsor-Investigator, Nghi Nguyen, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO17120310
Record Dates: First submitted 2018-01-23; First posted 2018-02-06 (Actual); Results first posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Cervical Cancer; Uterine Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms | interventions — fluciclovine F-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- 18F fluciclovine PET scan (Experimental): Subjects with recently biopsy-proven malignancy of the cervix or uterus undergo an 18F fluciclovine PET scan on a hybrid PET/MRI scanner after they have completed a standard-of-care F-18 FDG PET/CT study.
  Interventions: Drug: 18F fluciclovine; Device: 18F fluciclovine PET

INTERVENTIONS:
Drug: 18F fluciclovine — Each subject will receive one IV dose of 18F fluciclovine for PET scanning
  Other Names: Axumin
Device: 18F fluciclovine PET — Each subject will undergo one 18F fluciclovine PET scan on a hybrid PET/MRI scanner

SUMMARY:
18F Fluciclovine is a recently FDA- approved radiopharmaceutical for prostate cancer biochemical recurrence, which is only minimally eliminated by the kidneys and therefore the image interpretation is not affected by nonspecific urine activity in the ureters and bladder, which is advantageous for pelvic imaging. Recent literature suggests that Fluciclovine PET has diagnostic potential for a variety of solid tumors, thus, allowing new opportunities for noninvasive probing of glutamine metabolism and clinical use in patient management. Current literature indicates that amino acid transporters including that of glutamine are upregulated in endometrial and cervical cancer so that Fluciclovine PET may have clinical potentials. The hypothesis is that Fluciclovine PET provides better imaging properties and greater diagnostic confidence and accuracy than FDG PET does in pelvic malignancies.

Given the lack of current clinical data, a pilot study providing a direct comparison of Fluciclovine PET with FDG PET is warranted. The investigators seek to conduct a pilot study with 10 subjects to evaluate the clinical utility of Fluciclovine PET for staging of cervical cancer and endometrial cancer. This research will compare the diagnostic performance of the research Fluciclovine PET/MRI with the standard-of-care FDG PET/CT as an exploratory endpoint.

DETAILED DESCRIPTION:
Background:

Endometrial cancer arises from the inner lining of the uterus and is one of the most common malignancies in women, representing 3.6% of all new cancer cases in the US. It is estimated that there are more than 60,000 new cases of endometrial cancer and more than 10,000 people will die of this malignancy in 2016. It is most frequently diagnosed among women aged 55-64. Cervical cancer starts in the cervix, the lower part of the uterus. Its prevalence is lower compared with endometrial cancer thank to effective screening and early disease detection with the Pap smear. In 2016, it is estimated that there will be more than 12,000 new cases of cervical cancer and more than 4,000 patients will die of this disease in the US.

Positron Emission Tomography (PET) combined with Computed Tomography (CT) is an essential part of the workup for many malignancies. F-18 FDG PET/CT is currently the standard-of-care (SOC) PET/CT modality for staging and restaging of pelvic malignancies in women. But there are certain diagnostic limitations related to F-18 FDG because it is mainly eliminated by the kidneys and often interferes with the detection of cancer lesions, particularly in the abdominal and pelvic regions. On the other hand, the recently FDA approved F-18 Fluciclovine is only minimally eliminated by the kidneys and therefore the image interpretation is not affected by nonspecific urine activity in the ureters and bladder, which is advantageous for pelvic imaging. Recent literature suggests that Fluciclovine PET has diagnostic potential for a variety of solid tumors, thus, allowing new opportunities for noninvasive probing of glutamine metabolism and clinical use in patient management.

Current literature indicates that amino acid transporters including that of glutamine are upregulated in endometrial and cervical cancer so that Fluciclovine PET may have clinical potentials. The hypothesis is that Fluciclovine PET provides better imaging properties and greater diagnostic confidence and accuracy than FDG PET does in pelvic malignancies.

Given the lack of current clinical data, a pilot study providing a direct comparison of Fluciclovine PET with FDG PET is warranted.

Objective:

The investigators seek to conduct a pilot study to evaluate the clinical utility of Fluciclovine PET for staging of cervical cancer and endometrial cancer. This research will focus on pelvic imaging comparing the diagnostic performance of the research Fluciclovine PET/MRI with SOC FDG PET/CT as an exploratory endpoint. Dynamic PET imaging on a hybrid PET/MR scanner will provide valuable pharmacokinetic information that can be used to identify the optimal time window for the detection and characterization of the primary tumor and pelvic nodal disease. Additional abdominal imaging will allow for further correlation with FDG PET/CT in terms of nodal disease and distant metastasis detection. As previously demonstrated in prostate cancer, the Fluciclovine uptake can be heterogeneous which may have diagnostic and prognostic implications. Therefore, this pilot study will provide valuable information on potential Fluciclovine heterogeneity in cervical and uterine cancer. Textural heterogeneity of the primary will be compared between Fluciclovine and FDG PET. The initial experience gained with this pilot study will provide valuable insights into the pharmacokinetics and textural heterogeneity of Fluciclovine PET in cervical and uterine cancers, and presents the first data on the potential strengths and weaknesses of Fluciclovine PET/MR compared with FDG PET/CT.

1. The investigators hypothesize that Fluciclovine PET is non-inferior to FDG PET regarding detection of the primary tumor.
2. It is hypothesized that nodal disease staging is more accurate with Fluciclovine than with FDG PET because of the low level of nonspecific urinary bladder and ureter activity.
3. It is hypothesized that the dynamic uptake pattern of the primary lesion correlates with the tumor grading on histopathology.
4. It is hypothesized that textural heterogeneity is different between Fluciclovine and FDG PET.

Specific Aims:

* To study the pharmacokinetics of Fluciclovine PET in women with cervical and uterine cancers
* To characterize physiologic uptake pattern of the uterus and ovaries when these are not affected by tumor.
* To identify the optimal time window for the quantitative analysis of Fluciclovine primary and pelvic nodal disease
* To correlate the time-activity curve pattern of the primary lesion with histopathologic tumor grading
* To compare diagnostic performance of Fluciclovine PET and FDG PET
* To compare textural heterogeneity of the primary between Fluciclovine PET and FDG PET

Significance:

The initial experience gained with this pilot study will provide valuable insights into the pharmacokinetics, lesion detectability and textural heterogeneity of Fluciclovine PET in cervical cancer and uterine cancer. The study provides preliminary data on the potential strengths and weaknesses of Fluciclovine PET/MR compared with the SOC FDG PET/CT.

Fluciclovine PET may provide a significant improvement in the TNM staging compared with FDG PET as it is not affected by nonspecific urine activity in the ureters and bladder, which is a common diagnostic problem for FDG PET. By combining the excellent soft-tissue contrast of MRI with Fluciclovine PET, the hybrid PET/MR scanning could be a convenient and effective one-stop imaging procedure providing both pelvic TNM staging and whole-body M staging. Moreover, valuable prognostic information may be derived from Fluciclovine PET pharmacokinetics and heterogeneity assessment as well as multi-parametric PET/MR evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years and older
* Biopsy-proved cervical cancer or endometrial cancer within three months of study enrollment
* Standard-of-care (SOC) FDG PET/CT exam performed within 30 days of study enrollment

Exclusion Criteria:

* Female < 18 years old
* No history of cervical cancer or endometrial cancer
* Primary biopsy > 3 months of study enrollment
* Systemic therapy or radiation therapy initiated
* SOC FDG PET/CT exam performed > 30 days of study enrollment
* Therapeutic procedures (chemotherapy, radiation therapy) have been initiated
* Pregnancy or lactation
* Claustrophobia or inability to tolerate the imaging procedure on the PET/MR scanner
* Individual is not willing to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nghi C Nguyen, MD, PhD, Principal Investigator — Assistant Professor of Radiology
Locations (1):
- UPMC Presbyterian - MR Research Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available for this pilot study.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 18F Fluciclovine PET Scan
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 18F Fluciclovine PET Scan
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Lesion Metabolic Avidity
Description: Metabolic parameter of maximum standard-uptake-value (SUV) will be compared between research Fluciclovine PET and standard-of-care FDG PET to determine lesion metabolic avidity
Time Frame: Two weeks
Measure: Number; unit: g/dL
Arm/Group | 18F Fluciclovine PET Scan
Number analyzed (Participants) | 1
g/dL
  SUV of standard-of-care FDG | 21.5
  SUV of research Fluciclovine | 6.5

2. Secondary Outcome: Optimal Imaging Window
Description: The optimal time window for tumor detection (primary, nodal metastasis) relative to physiologic and benign structures will be determined based on time-activity curves of the Fluciclovine PET scan.
Time Frame: One hour
Population: Only one subject measured, so unable to determine optimal time window
Arm/Group | 18F Fluciclovine PET Scan
Number analyzed (Participants) | 0

3. Secondary Outcome: Fluciclovine PET Time-activity Curve Correlation With Histopathologic Tumor Grading
Description: The Fluciclovine time-activity curve of the primary tumor (time to peak, uptake intensity, and slope of washout) will be correlated with histopathologic tumor grading.
Time Frame: One hour
Population: Only one subject measured, so unable to determine correlation of time-activity-curve with histopathology.
Arm/Group | 18F Fluciclovine PET Scan
Number analyzed (Participants) | 0

4. Secondary Outcome: Textural Tumor Heterogeneity
Description: Parameters of textural tumor heterogeneity will be compared between Fluciclovine PET and FDG PET, using the open-access LIFEx software. The software allows for an automatic evaluation of more than 50 parameters for textural analyses and shows the result of the best parameters for tumor heterogeneity; however, no specific marker or measure of heterogeneity is be predefined in this process.
Time Frame: Two weeks
Population: Only one subject measured, so parameter output of software program would not be appropriate.
Arm/Group | 18F Fluciclovine PET Scan
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: One hour.
Arm/Group | 18F Fluciclovine PET Scan
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT03423082/Prot_SAP_001.pdf